CLINICAL TRIAL: NCT03707093
Title: A Study of CD137 Agonist ADG106 Administered Intravenously in Patients With Advanced or Metastatic Solid Tumors and/or Non-Hodgkin Lymphoma
Brief Title: Study of CD137 Agonist ADG106 With Advanced or Metastatic Solid Tumors and/or Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adagene Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADG106-1001
Record Dates: First submitted 2018-10-08; First posted 2018-10-16 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Solid Tumors, Non-Hodgkin Lymphoma
Keywords: Solid tumor; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADG106 Dose escalation (Experimental)
  Interventions: Drug: ADG106

INTERVENTIONS:
Drug: ADG106 — IV infusion over 60 minutes on Day 1 of each cycle, at doses of 0.03 mg/kg, 0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg,10 mg/kg or 300mg flat dose depending on cohort at enrollment.

SUMMARY:
This is a Phase 1, open-label, dose-escalation, multicenter study of ADG106 in subjects with advanced or metastatic solid tumors and/or relapsed/refractory non-Hodgkin lymphoma. ADG106 is a fully human ligand-blocking, agonistic anti-CD137 IgG4 mAb. It binds to the activated human T cells via a T cell receptor CD137. T cell is a kind of lymphocyte (a subtype of white blood cells) that protects bodies by eliminating tumor cells, and normal cells infected with viruses or bacteria. By binding to CD137, the study drug is expected to enhance the activity of activated T cells and thus stimulate a more intense immune attack to kill tumor cells. ADG106 is expected to enhance the activity of activated T cells.

The primary objective of the study is to assess safety and tolerability at increasing dose levels of single agent ADG106 in subjects with advanced or metastatic solid tumors and/or non Hodgkin lymphoma Secondary Objectives

* To characterize the pharmacokinetic (PK) profiles of ADG106
* To evaluate the immunogenicity of ADG106
* To evaluate the potential anti-tumor effect of ADG106 Exploratory Objective To identify the potential biomarkers of ADG106

ELIGIBILITY:
Inclusion Criteria

1. Male or female, 18 years of age or older at the time of consent.
2. Provide written informed consent.
3. Subjects with advanced and/or metastatic histologically or cytologically confirmed solid tumor and/or non-Hodgkin lymphoma who are refractory or relapsed from standard therapy and who have exhausted all available therapies.
4. Life expectancy of 12 weeks or greater.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. At least one measurable lesion per RECIST 1.1 for solid tumors and per Lugano Classification for non-Hodgkin lymphoma.
7. Adequate organ and bone marrow function
8. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within the 7 days prior to study drug administration.

Exclusion Criteria

1. Active central nervous system primary or secondary malignancies, active seizure disorder, spinal cord compression, or carcinomatous meningitis.
2. Any active autoimmune disease or documented history of autoimmune disease.
3. Infection of human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV), except for the following:
4. History of any non-infectious hepatitis (eg, alcohol or non-alcoholic steatohepatitis, drug-related or auto-immune hepatitis).
5. History of clinically significant cardiac disease.
6. Uncontrolled current illness.

8. WOCBP and sexually active fertile men with WOCBP partners who are unwilling or unable to use acceptable contraception method to avoid pregnancy.

9. Women who are pregnant at Screening or prior to study drug administration. 10. Women who are breastfeeding. 11. History of significant immune-mediated AE . 13. Systemic use of the following therapies within 28 days prior to the first dose of study drug, or longer.

14. Subjects who got either below treatment:

* Any previous anti-CD137 mAb (eg, utomilumab, urelumab) treatment.
* Subject who has received allogenic hematopoietic stem cell transplant or autologous stem cell transplanted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities | 2 Cycles (42 days)
Number of participants experiencing clinical and laboratory adverse events (AEs) | First dose to 28 days post last dose

SECONDARY OUTCOMES:
The area under the curve (AUC) of plasma concentration of drug | From first dose (Cycle 1 Day 1, each cycle is 21 days) until the last dose (up to 2 years)
Maximum concentration (Cmax) | From first dose (Cycle 1 Day 1, each cycle is 21 days) until the last dose (up to 2 years)
Time at which maximum concentration (Tmax) | From first dose (Cycle 1 Day 1, each cycle is 21 days) until the last dose (up to 2 years)
Lowest plasma concentration (C[trough]) | From first dose (Cycle 1 Day 1, each cycle is 21 days) until the last dose (up to 2 years)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Horizon Oncology Research, Lafayette, Indiana
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No